CLINICAL TRIAL: NCT05048134
Title: A Multi-center, Open-Label，Dose Escalation and Dose Expansion Phase I Study of HRS2300 Monotherapy or Combined With SHR-1316 or SHR-1701 or Trametinib or Almonertinib in Patients With Advanced Malignancies
Brief Title: A Phase I Study of HRS2300 or Combined With SHR-1316 or SHR-1701 or Trametinib or Almonertinib in Patients With Advanced Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor R&D strategy adjustment
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRS2300-I-101
Record Dates: First submitted 2021-08-31; First posted 2021-09-17 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Advanced Malignancies

STUDY DESIGN:
Intervention Model Description: HRS2300 monotherapy or combined with SHR-1316, SHR-1701, trametinib, and Almonertinib
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Treatment group A (Experimental)
  Interventions: Drug: HRS2300
- Treatment group B (Experimental)
  Interventions: Drug: HRS2300、 SHR-1316
- Treatment group C (Experimental)
  Interventions: Drug: HRS2300、SHR-1701
- Treatment group D (Experimental)
  Interventions: Drug: HRS2300、trametinib
- Treatment group E (Experimental)
  Interventions: Drug: HRS2300、Almonertinib

INTERVENTIONS:
Drug: HRS2300 — HRS2300 monotherapy
  Arms: Treatment group A
Drug: HRS2300、 SHR-1316 — HRS2300 combined with SHR-1316
  Arms: Treatment group B
Drug: HRS2300、SHR-1701 — HRS2300 combined with SHR-1701
  Arms: Treatment group C
Drug: HRS2300、trametinib — HRS2300 combined with trametinib
  Arms: Treatment group D
Drug: HRS2300、Almonertinib — HRS2300 combined with Almonertinib
  Arms: Treatment group E

SUMMARY:
The study is being conducted to evaluate the safety and tolerability of HRS2300 and combined with SHR-1316 or SHR-1701 or trametinib or Almonertinib.To Determine the maximum tolerated dose (MTD) and recommended Dose (RP2D) for HRS2300 monotherapy and combination therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years old，Male or female;
2. Patients with pathologically confirmed advanced solid tumors who did not respond to standard treatment, did not tolerate standard treatment, or were determined by the investigator to be unsuitable for standard treatment;
3. ECOG PS score of 0-1;
4. Life expectancy of ≥3 months;
5. Able and willing to provide a written informed consent.

Exclusion Criteria:

1. Receiving chemotherapy, targeted therapy, immunotherapy, radical radiotherapy or surgical treatment for less than 4 weeks before study therapy (excluding tyrosine kinase inhibitors or other small molecule targeted drugs < 2 weeks); Four weeks prior to the start of study treatment (patients who have entered the follow-up period measured by the time of last use of the experimental drug or device) were enrolled in another clinical study;
2. Drugs that affect the activity of metabolic enzyme CYP3A have been used in the past, and the eluting period from the end time to the first administration in this study is within 5 half-lives;
3. Patients with active TB within 1 year prior to the start of drug therapy or with a history of active TB infection more than 1 year prior to the start of drug therapy without proper treatment were studied;
4. Patients with other potential factors that may affect the study results or result in the premature discontinuation as determined by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-05-23 (Actual)

PRIMARY OUTCOMES:
Number of participants with Dose limited toxicity（DLT） | Cycle 1( 4 weeks- monotherapy；3 weeks -combination）
Number of participants with adverse events | up to 3 years; at least once per treatment cycle
Determine RP2D of HRS2300 monotherapy and combination in patients with advanced malignancy | through study completion，an average of 2 years
  Enrolled sequentially from the initial dose of the trial, each subject received only one dose of the study drug and no other dose. The first subject of each dose should complete the first administration and be observed for 7 days before the other two subjects can be enrolled. After the DLT observation period of the last subject in each dose group has ended, the next dose increment can be entered. At the end of the dose escalation phase, the dose closest to the estimated toxicity probability of the target was selected as the MTD . At the end of the dose escalation, the SMC determined the RP2D based on the previous data.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided